CLINICAL TRIAL: NCT05461079
Title: Association Between Anogenital Distance, Sperm Phenotype and Epigenetics in Infertile Men.
Brief Title: Sperm Phenotype and Differentially Methylated Regions
Acronym: Epigenetics
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Christian De Geyter, Prof. Dr.med., University of Basel
Other Study IDs: RME12072017
Record Dates: First submitted 2017-12-09; First posted 2022-07-15 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spermatozoa sorted with FACS according to two different staining methods: YoPro1 (apoptosis) and CMA3 (histone content). After sorting, we obtained four different groups: 1. YoPro1 positive and 2. YoPro1 negative, CMA3 positive and CMA3 negative. All sorted samples were stored frozen and sent for analysis of whole genome methylation status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subfertile men: 10 infertile men with shortened AGD (< 40 mm)
  Interventions: Diagnostic Test: obtention of up to three semen samples
- fertile semen donors: 10 fertile semen donors with normal AGD (>40 mm)
  Interventions: Diagnostic Test: obtention of up to three semen samples

INTERVENTIONS:
Diagnostic Test: obtention of up to three semen samples — sorting of spermatozoa with flow cytometry. In the presence of insufficient numbers of spermatozoa after sorting (<15 mill), up to three semen samples will be collected.
  Other Names: conventional semen analysis followed by sorting

SUMMARY:
Testicular dysgenesis syndrome (TDS) is known to cause epigenetic abnormalities in spermatozoa. Anogenital distance (AGD) is considered to be a suitable clinical marker of TDS, but the direct link between AGD and epigenetic abnormalities is still missing.

Infertile men (n=10) presenting with shortened AGD and a control group of normal semen donors (n=10) with normal AGD will then be asked to provide one semen sample each. Using a flow cytometer and sorter (FACS) their spermatozoa will be sorted into populations of spermatozoa with/without DNA fragmentation or with/without chromatin decondensation. These sorted populations of spermatozoa will then be examined for differences in epigenetic imprinting differences using whole genome expression analysis. Whereas the sorting of spermatozoa will be carried out in Basel, the epigenetic analysis will be carried at the University of Geneva.

DETAILED DESCRIPTION:
A subset of 10 men with shortened AGD (together with a control group of 10 fertile donors with normal AGD) will be asked to provide up to three semen samples, each of which then will be sorted with FACS into subpopulations with/without DNA fragmentation and into subpopulations with/without chromatin decondensation.

Spermatozoa with fragmented DNA will be separated through FACS-sorting of spermatozoa with intact DNA using the YoPro 1-dye, which has been shown to correlate significantly with the degree of DNA fragmentation in the nuclei of sperm.

In addition, spermatozoa with abnormal chromatin remodelling will be separated through sorting from spermatozoa with condensed chromatin using the fluorochrome chromomycin A3 (CMA3), which competes for protamin for binding to the minor groove of DNA thereby correlating with the persistence of histones in the sperm nuclei. Pilot experiments have demonstrated the highly significant and close correlation of CMA3 with anilin blue staining. Anilin blue staining is not suitable for the sorting experiment, because it requires fixation of the spermatozoa. Sorting based on CMA3 can be carried out with living spermatozoa.

The sorted and anonymized samples will then be sent frozen in dry ice to a laboratory at the University of Geneva for the assessment of differences in the epigenetic imprinting of the DNA using whole genome expression studies.

ELIGIBILITY:
Inclusion Criteria:

* infertile men with known anogenital distance

Exclusion Criteria:

* sperm concentration must be more than 15 million/ml to allow appropriate sorting with flow cytometry...

Ages: 20 Years to 55 Years | Sex: Male
Age Groups: Adult
Study Population: Both the 10 infertile men with shortened AGD and the fertile control men (semen donors) will be recruited and examined in the infertility consultation of the Clinic of Gyn. Endocrinology and Reproductive Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
anogenital distance and epigenetics | 6 months
  number of differentially methylated transposable regulatory sequences in the genome of sorted spermatozoa.

SECONDARY OUTCOMES:
sperm phenotype 1 | 6 months
  based on conventional semen analysis: concentration of spermatozoa (in mill/ml).
sperm phenotype 2 | 6 months
  based on conventional semen analysis: progressive motility (in %).
sperm phenotype 3 | 6 months
  based on conventional semen analysis: normal morphology (in %), staining).
sperm phenotype 4 | 6 months
  chromatin decondensation (as given by % of CMA3 staining).
sperm phenotype 5 | 6 months
  DNA fragmentation (% of YoPro 1-staining).

CONTACTS AND LOCATIONS:
Locations (1):
- Christian De Geyter, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No